CLINICAL TRIAL: NCT00674544
Title: Influence of a Lifestyle Intervention in Preschool Children on Physiological and Psychological Parameters (Ballabeina)
Brief Title: Influence of a Lifestyle Intervention in Preschool Children on Physiological and Psychological Parameters
Acronym: Ballabeina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University of Basel (Other)
Responsible Party: Dr. Jardena Puder, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3200BO-116837
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2009-04

CONDITIONS: Obesity
Keywords: childhood; children; obesity; physical activity; nutrition; fitness; family
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No intervention, regular kindergarten program
- Intervention group (Experimental): Kindergarten and homebased increases in physical activity, healthy nutrition, sleep duration and decrease in media use: Involvement of parents and siblings
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Kindergarten and homebased increases in physical activity, healthy nutrition, sleep duration and decrease in media use: Involvement of parents and siblings
  Arms: Intervention group

SUMMARY:
Childhood obesity and low fitness tracks into adulthood and carries significant co-morbidities. The investigators test the hypothesis that a multidisciplinary multilevel lifestyle intervention in preschool children in the French and German speaking part of Switzerland during one school-year results in a smaller increase in body mass index (BMI) and a larger increase in aerobic fitness.

DETAILED DESCRIPTION:
We will assess the effect of this multidisciplinary intervention in a multicenter cluster randomized controlled trial including a total of 40 kindergarten classes in the French (canton Vaud) and in the German (canton St. Gallen) speaking part of Switzerland. Health promoters, trained in physical education, will receive further postgraduate training (in nutrition, education, psychology) and will then in reward teach several kindergarten teachers hands-on. These trained health promoters will intervene on the level of the kindergarten teacher, the parents, the local community and also on the level of the children following a professional pre-specified curriculum in the kindergarten that focuses primarily on physical activity, healthy nutrition, media use and sleep duration. The curriculum also includes information evenings, workshops and fun weekly homework packages. Special attention will be paid to establish a curriculum that reaches also socio-cultural high risk groups living in Switzerland. Measurements will be performed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy kindergarten children

Exclusion Criteria:

* Children with severe chronic disease (restricting physical activity)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 650 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
BMI and aerobic fitness | 1 schoolyear

SECONDARY OUTCOMES:
total and central body fatness | 1 schoolyear
motor abilities | 1 schoolyear
physical activity | 1 schoolyear
Media use | 1 schoolyear
Nutritional behavior and food intake | 1 schoolyear
Cognition tests | 1 schoolyear
Health-related quality of life, presence of hyperactivity | 1 schoolyear

CONTACTS AND LOCATIONS:
Overall Officials: Jardena J Puder, MD, Principal Investigator — University of Lausanne
Locations (1):
- Service of Endocrinology, Diabetes and Metabolism; University of Lausanne, Lausanne, Switzerland

REFERENCES:
- [Derived] Puder JJ, Marques-Vidal P, Schindler C, Zahner L, Niederer I, Burgi F, Ebenegger V, Nydegger A, Kriemler S. Effect of multidimensional lifestyle intervention on fitness and adiposity in predominantly migrant preschool children (Ballabeina): cluster randomised controlled trial. BMJ. 2011 Oct 13;343:d6195. doi: 10.1136/bmj.d6195. PMID 21998346
- [Derived] Niederer I, Kriemler S, Gut J, Hartmann T, Schindler C, Barral J, Puder JJ. Relationship of aerobic fitness and motor skills with memory and attention in preschoolers (Ballabeina): a cross-sectional and longitudinal study. BMC Pediatr. 2011 May 11;11:34. doi: 10.1186/1471-2431-11-34. PMID 21569343
- [Derived] Burgi F, Meyer U, Granacher U, Schindler C, Marques-Vidal P, Kriemler S, Puder JJ. Relationship of physical activity with motor skills, aerobic fitness and body fat in preschool children: a cross-sectional and longitudinal study (Ballabeina). Int J Obes (Lond). 2011 Jul;35(7):937-44. doi: 10.1038/ijo.2011.54. Epub 2011 Mar 29. PMID 21448128
- [Derived] Burgi F, Meyer U, Niederer I, Ebenegger V, Marques-Vidal P, Granacher U, Kriemler S, Puder JJ. Socio-cultural determinants of adiposity and physical activity in preschool children: a cross-sectional study. BMC Public Health. 2010 Nov 26;10:733. doi: 10.1186/1471-2458-10-733. PMID 21110865
- [Derived] Niederer I, Kriemler S, Zahner L, Burgi F, Ebenegger V, Hartmann T, Meyer U, Schindler C, Nydegger A, Marques-Vidal P, Puder JJ. Influence of a lifestyle intervention in preschool children on physiological and psychological parameters (Ballabeina): study design of a cluster randomized controlled trial. BMC Public Health. 2009 Mar 31;9:94. doi: 10.1186/1471-2458-9-94. PMID 19335890